CLINICAL TRIAL: NCT04284371
Title: The Prevalence of Liver Steatosis, Steatohepatitis, Fibrosis, and Hemosiderosis in Overweight and Obese US Military Dependent Pediatric Patients Using MR Elastography and Quantitative MRI
Brief Title: The Prevalence of Nonalcoholic Fatty Liver Disease (NAFLD) Pediatric Patients
Status: Terminated | Type: Observational
Why Stopped: lack of funding - no results to report
Sponsor: The Geneva Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: C.2016.01
Record Dates: First submitted 2019-11-25; First posted 2020-02-25 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Steatohepatitis, Nonalcoholic; Hemosiderosis; Overweight Adolescents; Obesity, Childhood; Liver Steatosis
Keywords: Liver Steatosis; Overweight Adolescents
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hemosiderosis; Pediatric Obesity; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of liver steatosis, steatohepatitis, fibrosis, and hemosiderosis in overweight and obese US Military dependent pediatric patients using MR Elastography and Quantitative MRI

DETAILED DESCRIPTION:
The purpose of this prospective study is to determine the prevalence NAFLD and of factors that have been associated with the diagnosis of fatty liver disease in overweight and obese children and adolescents and to determine the effectiveness of an intervention. In order to do this, we will also compare laboratory values and the ability/feasibility of new magnetic resonance technologies to first detect fatty liver disease and then to detect a difference in liver health between pediatric patients with a normal BMI and those with a BMI ≥85%. This study will consist of two phases and a reproducibility arm involving 19 voluntary subjects from Phase 1 and the control group.

Phase I:

Aim 1: To determine the prevalence and relative risk of liver fibrosis, steatosis, steatohepatitis and hemosiderosis in overweight and obese US Military dependents between ages 10 and 17 compared with normal weight controls using specialized MRI (LMS).

Aim 2: To compare results between MRI-LMS and MRE and to determine feasibility of one versus the other technology.

Aim 3: To compare liver health of controls and overweight/obese subjects to determine if there is a difference between groups.

Aim 4: To test for various biomarkers that have been shown to have an association with NASH

Phase II:

Aim 1: To evaluate the effectiveness of a nine month intervention consisting of diet and exercise education on the maintenance or reduction of liver steatosis, steatohepatitis, and fibrosis.

Aim 2: To establish whether early imaging can predict short-term clinical outcomes (eg development of pre-diabetes, worsening NAFLD, development of NASH, or a change in liver stiffness or fibrosis as measured by MRE and LMS, respectively).

Reproducibility Arm Aim 1: To evaluate the consistency of the LMS/MRE data.

ELIGIBILITY:
Inclusion Criteria:

1. DEERS eligible patients from the San Antonio Military Medical Center Healthy Habits clinic and pediatric endocrine, pediatric gastroenterology, adolescent, and general pediatric clinics, as well as from Wilford Hall's pediatric clinic.
2. Overweight (BMI > 85% and < (Control group) Normal BMI for age and gender (BMI <85%) 95% for age and gender) or obese (BMI >/= 95% for age and gender)
3. 10 - 17 years old
4. Cognitively able to understand and provide written informed assent
5. Written informed consent from parent or legal guardian

Exclusion criteria:

1. Current or prior history of liver disease (to include chronic hepatitis B or C, hemochromatosis, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, HIV, biliary atresia, or Caroli/choledochal disease), or other known liver disease.
2. Pregnancy (self-reported or through positive beta HCG test during study)
3. Current use of hepatotoxic medications associated with liver disease/failure (antifungals, methotrexate, valproic acid)
4. Carrying an implantable active medical device such as a pacemaker, vagal nerve stimulator, defibrillator, or non-MRI compatible cochlear implant.
5. Previous claustrophobia/anxiety with MRI scanner or developmental delays that may result in failed MRI scan (e.g.autism, anxiety disorder)
6. Any alcohol use
7. Predicted family PCS/loss of benefits in the next 9 months (Phase II only)

Ages: 10 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Military dependent population male and females age 10-17 years of age
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
LiverMultiScan (LMS) | 2 years
  LMS Imagery will be used to for observance of the prevalence of liver fibrosis, steatosis, steatohepatitis and hemosiderosis on LMS in overweight and obese US Military dependents between ages 10 and 17
MRE | 24
  MRE imagery will be used as a comparison to the LMS imagery to help determine Liver stiffness as measured by MRE overweight and obese US Military dependents between ages 10 and 17after a 9 month intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christian Carlosn, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States